CLINICAL TRIAL: NCT06288971
Title: Personalized Innovative Intervention Pathways to Promote Executive Function in Children With Cerebral Palsy
Brief Title: Personalized Innovative Intervention Pathways to Promote EF in Children With CP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: University of Pisa (Other); University of Florence (Other); Anastasis Società Cooperativa Sociale (Unknown)
Responsible Party: Principal Investigator, Giuseppina Sgandurra, MD, PhD, IRCCS Fondazione Stella Maris
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRCCS FSM
Record Dates: First submitted 2024-02-26; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Executive Functions in Cerebral Palsy
Keywords: Cerebral Palsy; Executive Function; Neuropsychological Evaluation; Neuropsychological Rehabilitation; Educational Robotics; Game-based System; Instrumental School Learning Skills
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Children with impairment in EF and in visuo-spatial abilities (Experimental): Children aged 5 to 13 years old with a diagnosis of Cerebral Palsy, with EF impairment and visuo-spatial difficulties
  Interventions: Other: Self-adaption web-based software for the rehabilitation of EF and visuo-spatial abilities
- Children with impairment in EF and in specific cognitive processes underlying academic skills (Experimental): Children aged 5 to 13 years old with a diagnosis of Cerebral Palsy, with impairment in EF and in specific cognitive processes underlying academic skills
  Interventions: Other: Tele-rehabilitation of EF and specific cognitive processes underlying academic skills
- Children with impairment in EF and in motor planning (Experimental): Children aged 5 to 13 years old with a diagnosis of Cerebral Palsy, with impairment in EF and in motor planning
  Interventions: Other: Game-based tools for the rehabilitation of EF and motor planning
- Typically developing children (No Intervention): Children aged 5 to 13 years old with no clinically documented disorders.

INTERVENTIONS:
Other: Self-adaption web-based software for the rehabilitation of EF and visuo-spatial abilities — - Self-adaption web-based software integrated with neuropsychomotor activities in small groups to strengthen EF. The training will take place bi-weekly, for 3 months, for approximately 60 minutes per meeting. For the intervention will be used the Bee-bot, a robot to be programmed to achieve objectives set in space, allows to stimulate navigation, visuospatial working memory and planning skills (the activities will be taken from those already used in our previous studies in children with typical development and BES (Di Lieto et al., 2020)).
  Arms: Children with impairment in EF and in visuo-spatial abilities
Other: Tele-rehabilitation of EF and specific cognitive processes underlying academic skills — - Tele-rehabilitation intervention on FE (RuntheRAN and MemoRAN). The training will be conducted at home, with periodic meetings with the clinician, for 3 months, for approximately 4/5 days a week for approximately 30/40 minutes per day. An adult (e.g. a family member) will support the child in the treatment and ensure that the exercises are carried out adequately at home. One of the following tele-rehabilitation software will be used: RuntheRAN (RidiNet, Coopertiva Sociale Anastasis), a software that aims to strengthen the prerequisites of reading by requiring the timed and progressively faster naming of colour matrices or black and white figures. MemoRAN (RidiNet, Cooperativa Sociale Anastasis), which involves rapid naming exercises of stimuli (figures and colors) presented in matrices, within tasks that require inhibition, cognitive flexibility and updating in working memory.
  Arms: Children with impairment in EF and in specific cognitive processes underlying academic skills
Other: Game-based tools for the rehabilitation of EF and motor planning — - MondoELLI intervention (Cooperativa Sociale Anastasis) integrated with neuropsychomotor activities. The game-based app involves activities in small groups to strengthen various components of EF (interference control, inhibition, working memory, flexibility). The activities are organized with increasing difficulty, according to the self-adaptive algorithm, and within a narrative context.
  Arms: Children with impairment in EF and in motor planning

SUMMARY:
Cerebral palsy (CP) is an umbrella term, covering a group of disorders of movement and posture. It is now accepted that CP represents much more than a disorder of movements considering the frequent association with a broad range of impairments, including cognitive impairments. In general, multiple clinical characteristics that define and determine different functional profiles. Several studies on children with unilateral and bilateral CP have been shown that, despite the overall preserved intellectual functioning, there are specific neuropsychological impairments distinguishing the two forms, including deficits in different Executive Functions (EF) components. Executive Functions (EFs) represent a complex cognitive domain consisting of a set of top-down functions essential for adaptive goal-directed behaviour, allowing to formulate, plan, and organise ideas, cope with challenges and novelties, resist temptations and stay focused. EF represents general domain abilities transversal to several cognitive processes and underling different daily life activities and school learning skills. Empowering EF becomes therefore crucial in children with CP both to strengthen specific functional EF weaknesses and to achieve far transfer effects on other compromised domains, such as motor planning, academic skills,and/or visuospatial processing. To pursue this, the EF training needs to be integrated into the complex and multidisciplinary care context promoting innovative intervention methodologies based on scientific evidence. Recent researches and clinical practice, carried out in our Institute, supports the effectiveness of innovative interventions on EF using new technologies in typical and atypical development, such as Self-adapting web based softwares, Game-based tools or Educational Robotics. Literature suggests these technologies allow to promote timely intervention within a user-friendly context, while respecting the key criteria of evidence-based neuropsychological rehabilitation, both reducing hospitalisation times and supporting interest and motivation for participation. The primary aim of this study is to evaluate the applicability of technological intervention integrated with psychomotor activities to promote EF and then secondary to measure the effect on the functional profile of children with CP, including motor planning, visuo-spatial processing and learning skills, evaluating both short-term (T2) and long-term changes (T3).

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is an umbrella term, covering a group of permanent disorders of movement and posture development, causing activity limitation. It is now widely accepted that CP motor disorders are frequently associated with a broad range of functional impairments, including cognitive and neuropsychological functions. The presence of epilepsy, premature birth, low birth weight, reduced fetal growth, lesion characteristics and severe gross motor impairment are significant risk factors for cognitive deficit development. Due to the great heterogeneity of the clinical pictures, which depend on the extent, magnitude and timing of the lesion, it is possible to distinguish different forms of CP (International Classification of 2013): spastic forms (approx. 90% of total cases), dyskinetic and ataxic forms. Research indicates a better functional outcome in children with spastic hemiplegia and diplegia compared to those with tetraplegic and ataxic CP, where severe intellectual deficits are more commonly reported, although significant challenges in the standardized assessment of these children are due to more severe motor and oro-motor impairment (Ballester-Plane et al., 2018). A more substantial number of studies have been conducted on children with spastic hemiplegia and diplegia, revealing that, despite overall preserved intellectual functioning, there are specific neuropsychological impairments distinguishing unilateral and bilateral CP. Deficits in different Executive functions (EF) components, playing an important role in behaviour regulation, problem solving, social abilities and the successful completion of everyday activities, are also often reported in literature. One of the reference theoretical models for EFs is the one proposed by Adele Diamond who, starting from Miyake's fractional model, described EFs as made up of three main components (inhibitory control, working memory and cognitive flexibility) which allow the structuring of higher order EFs (reasoning, planning and problem solving). Several studies have identified a close association between EF and other domains considering such processes as transversal to several cognitive and motor functions, also underlying different daily life activities and school learning skills (such as mathematics, reading or writing). The role of specific training on EF becomes crucial in children with CP both to strengthen specific EF weaknesses and to achieve generalised benefits in other compromised domains, such as motor planning, visuospatial processing or academic achievements. To pursue this, the training needs to be integrated into the complex and multidisciplinary care context in which the child with neuromotor disorder is already placed. Recent years have seen the spread of innovative rehabilitation methods, such as Self-adapting web-based software, Game-based systems or Educational Robotics. Literature suggests these technologies have the advantage of intervening in a timely manner, within a home-based context , while following the the key criteria of evidence-based neuropsychological rehabilitation (intensity, self-adaptivity of the exercise and planning fun, enjoyable and motivating activities). In particular, Self-adapting web-based software improving the difficulties of the activities delivered according to the children's performance is used in several neurodevelopmental disorders for the treatment of motor, cognitive, learning and language impairments (e.g. Capodieci et al., 2022).

Game-based tools facilitate meaningful learning, through serious game activities exploiting playful elements and delivering continuous feedback on children's performance. As its video-game nature, the difficulty is adapted to the children' skills and rises progressively according to the learning aims. Educational Robotic (ER) refers to a learning approach requiring children to design, assemble, and program robots through play and hands-on activities. Robot programming may be a tool to increase problem solving skills, cognitive flexibility and inhibition in both typical and atypical development (Di Lieto et al., 2019 and 2020). It is possible to profitably use all of these tools in children with Cerebral Palsy (CP), considering their neuropsychological and motor function impairments.

The aim of this study is to evaluate the applicability and effect of technological intervention integrated with psychomotor activities to promote EF and secondary the impact on academic skills and motor planning in children with CP, evaluating both short-term (T2) and long-term changes (T3). More specific outcomes will be:

* To verify the feasibility of using new intervention technologies, adopting intensive and self-adaptive methodologies and encouraging interaction and learning between peers.
* To build three personalised intervention protocols based on the different neuropsychological profiles.
* To analyse the effect of such intervention on the EF directly targeted
* To evaluate the generalised effect of the EF intervention on other domains, such as academic skills, visuo-spatial processing and motor planning.

Both short-term (T2) and long-term (T3) changes will be considered.

The attribution to the following treatment paths will not be completely randomised, because based on specific children rehabilitation needs, both considering age and neuropsychological profile:

* Educational Robotics integrated with psychomotor activities (ERi) in small groups to strengthen EF. The training will take place bi-weekly, for 3 months, for approximately 60 minutes per meeting. For Educational Robotics will be used the Bee-bot, a robot bee-like to program its movement using some directional buttons on the back in order to achieve and reach objectives set in space, therefore allowing to stimulate navigation, visuospatial working memory and planning skills (the activities will be taken from those already used in our previous studies in children with typical development and BES (Di Lieto et al., 2020).
* Self-adaptive web-based software on EF (RuntheRAN and MemoRAN; https://www.anastasis.it). The training will be conducted at home, for 3 months, for approximately 4/5 days a week for approximately 30/40 minutes per day. An adult (e.g. a family member) will support the child in the treatment and ensure that the exercises are carried out adequately at home. The clinician can monitor and control the intervention progress, also intervening manually on the auto-adaptation, both in online sessions and offline. For the intervention will be used: RuntheRAN (RidiNet, Coopertiva Anastasis), a software that aims to strengthen the prerequisites of reading by requiring the timed and progressively faster naming of colour matrices or black and white figures; MemoRAN (RidiNet, Cooperativa Anastasis), which involves rapid naming exercises of stimuli (figures and colours) presented in matrices, within tasks that require inhibition, cognitive flexibility and updating in working memory.
* The ELLI's WORLD (https://www.anastasis.it/il-mondo-degli-elli/) integrated with psychomotor activities. The game-based app involves activities in small groups to promote various components of EF (interference control, inhibition, working memory, flexibility). The activities are organised with increasing difficulty, according to the self-adaptive algorithm, and within a narrative context.

The clinical sample will be evaluated at different times during the study period: T1, T2, T3.

The study involves 3 functional assessments: pre-training (T1), after 3 months from T1 assessment for post-training (T2) and after 6 months from T2 assessment for follow-up (T3).

The short-term effect of the treatment will be evaluated by comparing pre- post assessment and the degree of improvement during the training (Percentage of Nonoverlapping Data, https://ktarlow.com/stats/pnd). The long-term effect will be analysed 6 months after the end of the intervention by comparing the performances post intervention with those at the follow-up.

ELIGIBILITY:
Children with Cerebral Palsy:

Inclusion Criteria:

* Children with confirmed diagnosis of CP
* Ages from 5 to 13 years old
* At least one cognitive index > 85 at WPPSI-IV or WISC-IV
* Functional weakness in EF

Exclusion Criteria:

* Severe comorbidities and/or severe cognitive disability

For Typically developing children:

* Ages from 5 to 13 years old
* No documented clinically relevant disorders

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
changes in score of inhibition subtest at the NEPSY-II | 1-36 months
  In the study the investigators will assess the Inhibition subtest at the NEPSY-II (Urgesi et al., 2011). that valuates the ability to inhibit automatic responses in favour of novel responses and to switch between response types. It is divided into three conditions: naming, inhibition and switching. Both accuracy and speed are obtained for each condition, with standardised score range from 1 to 19. Higher scores revealed better performances.

SECONDARY OUTCOMES:
changes in score of the sustained attention subtest at the Leiter-3 | 1-36 months
  In this study, the investigators will use the Sustained Attention subtest at the Leiter International Performance Scale (Leiter-3) (Roid et al., 2013), which assesses visual attention and consists of repetitive barrage tasks to be performed in a predefined time. The number of correctly selected target elements are recorded. Raw scores range from 0 to 217, while standardised score range from 1 to19. Higher scores revealed better performances.
changes in score of Developmental Test of Visual-Motor Integration (VMI) | 1-36 months
  VMI (Beery & Buktenica, 2000) is a paper-pencil test used to determine the level of integration between visual and motor systems. The child will be asked to copy different geometric forms shown on the paper within a certain time frame. The number of figures correctly reproduced is recorded and then converted in standardized scores. Raw scores range from 0 to 27. Higher scores reveal a better performance.
changes in score of MOXO-continuous performance test | 1-36 months
  MOXO evaluates sustained attention and is provided via a computer. The test requires the child to sustain attention over a continuous stream of stimuli (visual or auditory) and to respond to a specific target stimulus. Four scales are extracted and converted in z scores: attentiveness, timeliness, impulsiveness, hyper-reactivity. Higher scores reveal a better performance.
changes in score of Corsi block-tapping subtest at the BVS-corsi | 1-36 months
  The Corsi block-tapping subtest at the BVS-corsi (Mammarella et al., 2008) evaluates visuo-spatial short-term and working memory. The child is asked to retrieve a sequence previously seen by the examiner by tapping blocks with the preferred finger following the same order for the forward condition or reversing the order for the backward condition. The length of the last sequence correctly retrieved is recorded as the span, ranging from 3 to 8 in the forward condition and from 2 to 7 in the backward. Higher span reveals better performance.
changes in score of Behaviour Rating Inventory of Executive Function (BRIEF-P/2) for parents | 1-36 months
  BRIEF-P/2 (Gerard et al, 2016) is a questionnaire filled in by the parents/legal guardians and dives into everyday behaviour associated with specific domains of the executive functions (i.e., mental processes that enable us to plan, focus attention, remember instructions). Parents rate items (e.g., "does not think before doing") on a three-point scale ranging from 1 (never) to 3 (often). In the BRIEF 2 version, 9 scales are then extracted and converted in T scores: inhibition (ranging 8-24), self-monitoring (ranging 4-12), shift (ranging 8-24), emotional regulation (ranging 8-24), initiate (ranging 5-15), working memory (ranging 8-24), plan/organize (ranging 8-24), task monitoring (ranging 5-15), material organization (ranging 6-18); in the BRIEF P version, 5 scales are then extracted and converted in T scores: inhibition (ranging 16-48), shift (ranging 10-30), emotional regulation (ranging 10-30), working memory (ranging 17-51), plan/organize (ranging 10-30).
changes in score of RAN (rapid automatized naming) subtest at the rapid automatized naming and visual search of colours, figures and numbers test. | 1-36 months
  In the study the investigators will assess the subtest rapid visual naming (RAN) at the rapid automatized naming and visual search of colours, figures and numbers test (De Luca et al., 2005): the task consists in naming aloud all the stimuli contained in each matrix (colours, figures and numbers). For both tests time and number of errors are measured.
changes in score of reading and text comprehension task at the ALCE | 1-36 months
  ALCE (Bonifacci et al., 2014) is a test for the evaluation of learning difficulties and for the evaluation of reading and comprehension skills. In the study the investigators will assess two subtests:
  * Reading of the passage (in which the child is asked to read a passage, considering speed and correctness).
  * Reading comprehension (in which the comprehension skills of a read text are tested).
changes in score of reading and writing task at the DDE-2 | 1-36 months
  The battery for the Evaluation of Dyslexia and Developmental Dysortography-2 (DDE-2) (Sartori et al., 2007) is a test to evaluate reading and writing skills in children. In the study the investigators will assess two subtests:
  * Test 2 and 3 (reading words and non-words, in which the child is asked to read aloud as quickly and as accurately as possible 4 lists of 28 concrete and abstract words with high or low frequency and 3 lists of 16 non-words, in line with the phonotactic and phonographic rules of the Italian language).
  * Test 6 and 7 (writing words and non-words under dictation, in which the child is asked to write 48 concrete and abstract words with high or low frequency and 24 non-words).
changes in score of digit span forwards and backwards subtest at the BVN 5-11 and BVN 12-18 | 1-36 months
  In the study the investigators will assess the subtests digit span forwards and backwards at the BVN 5-11 (Bisiacchi et al., 2005) and BVN 12-18 (Gugliotta et al., 2009) for assess short-term and working memory, the child is asked to repeat the numbers spoken by the examiner following the same order for the forward condition or reversing the order for the backward condition. The length of the last sequence correctly retrieved is recorded as the span, ranging from 3 to 9 in the forward condition and from 2 to 8 in the backward. Higher span reveals better performance.
changes in score of Go/No-Go and N-back 1 subtest at the teleFE | 1-36 months
  TeleFE (Cooperativa Sociale Anastasis) is a web platform for the multidimensional assessment of Executive Functions in developmental ages from 6 to 13 years. In the study the investigators will assess three subtests:
  * In the go/no-go subtest children are asked to press a button when they see only the target stimulus between distracting stimuli that appear on the screen.
  * In subtest n-back 1, children are asked to remember the same item as the previous one within a string of stimuli that appear on the screen.
  Both accuracy and speed are scored for each subtest, with percentile score. Higher scores revealed better performances.
changes in score of verbal fluency subtest at the NEPSY-II | 1-36 months
  In the study the investigators will assess the Verbal Fluency Subtest at the NEPSY-II (Urgesi et al., 2011), in which the child is asked to generate in one minutes as many words as possible from a given category (animals, food and drinks) or with an initial phoneme (F and S). The test evaluates lexical access and total number of correctly generated word is scored for both the semantic and the phonological condition. The standardised score range is from 1 to 19. Higher scores revealed better performances.
changes in score of Test of Visual Perception and Visuo-motor Integration (TPV) | 1-36 months
  TPV (Hammill, 1994) is a test for the evaluation of visuo-perceptual and visuo-motor integration skills. In the study the investigators will assess the subtests:
  * Copying\ reproduction Subtest: the child sees figures that he must copy
  * Visual\motor speed: the child is asked to draw distinctive designs inside the target figures.
  * Hand-eye coordination: the child is asked to draw some lines inside bands of different widths.
  * Spatial relationships: the child is asked to connect some dots to reproduce the target figure.
  From these four subtests, the visual-motor integration score can be calculated and converted into a percentile score. Higher scores revealed better performances.
changes in score of Praxic and Motor Coordination Skills-2nd Edition (APCM-2) | 1-36 months
  APCM-2 (Sabbadini, 2015) aims to assess motor and praxis skills in children aged between 2-8 years, with age goup-specific performance tests.APCM-2 enables the early identification of deficits in motor-praxic coordination. The obtained scores facilitate a comprehensive assessment of each case, delineating the functional profile by calculating the deviation from the normative mean and referencing percentile values (5°, 10°, 25°). This approach aids in pinpointing specific functions for each scale, ranging from the most intact to the most impaired.
changes in score of Movement Assessment Battery for Children - Second Edition (Movement ABC-2) | 1-36 months
  Movement ABC-2 (Henderson, 2013) evaluates movement difficulties in 3 to 16 years children and adolescents. This assessment battery examines motor difficulties in children and adolescents aged 3 to 16 years. Tasks are categorized by age group and distributed across three sections: manual dexterity, aiming and catching, and balance. Scores are presented in standard scores and percentiles, with interpretation facilitated by a traffic light system. A green light signifies typical motor performance (scores above the 15th percentile), a yellow light indicates a risk for motor impairment (scores between the 5th and 15th percentile), and a red light identifies a significant motor function impairment (scores below the 5th percentile).
changes in score of Synthetic scale for the evaluation of writing in developmental age (BHK test) | 1-36 months
  The BHK test (Hamstra-Bletz et al., 2010) evaluates developmental dysgraphia, both the poor quality of the graphic sign (morphological analysis) and the disfluency (speed in the production of graphemes). Both accuracy and speed are evaluated with a z score and a percentile score, respectively. Higher scores reveal better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppina Sgandurra, MD, PhD, Principal Investigator — IRCCS Fondazione Stella Maris
Locations (1):
- IRCCS Fondazione Stella Maris, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fluss J, Lidzba K. Cognitive and academic profiles in children with cerebral palsy: A narrative review. Ann Phys Rehabil Med. 2020 Oct;63(5):447-456. doi: 10.1016/j.rehab.2020.01.005. Epub 2020 Feb 19. PMID 32087307
- [Background] Zoccolotti P, Cantagallo A, De Luca M, Guariglia C, Serino A, Trojano L. Selective and integrated rehabilitation programs for disturbances of visual/spatial attention and executive function after brain damage: a neuropsychological evidence-based review. Eur J Phys Rehabil Med. 2011 Mar;47(1):123-47. PMID 21448124
- [Background] Diamond A, Ling DS. Conclusions about interventions, programs, and approaches for improving executive functions that appear justified and those that, despite much hype, do not. Dev Cogn Neurosci. 2016 Apr;18:34-48. doi: 10.1016/j.dcn.2015.11.005. Epub 2015 Dec 7. PMID 26749076
- [Background] Di Lieto MC, Castro E, Pecini C, Inguaggiato E, Cecchi F, Dario P, Cioni G, Sgandurra G. Improving Executive Functions at School in Children With Special Needs by Educational Robotics. Front Psychol. 2020 Jan 9;10:2813. doi: 10.3389/fpsyg.2019.02813. eCollection 2019. PMID 31998169
- [Background] Pecini C, Spoglianti S, Bonetti S, Di Lieto MC, Guaran F, Martinelli A, Gasperini F, Cristofani P, Casalini C, Mazzotti S, Salvadorini R, Bargagna S, Palladino P, Cismondo D, Verga A, Zorzi C, Brizzolara D, Vio C, Chilosi AM. Training RAN or reading? A telerehabilitation study on developmental dyslexia. Dyslexia. 2019 Aug;25(3):318-331. doi: 10.1002/dys.1619. Epub 2019 May 23. PMID 31124262
- [Background] Diamond A. Executive functions. Annu Rev Psychol. 2013;64:135-68. doi: 10.1146/annurev-psych-113011-143750. Epub 2012 Sep 27. PMID 23020641
- [Background] Di Lieto MC, Brovedani P, Pecini C, Chilosi AM, Belmonti V, Fabbro F, Urgesi C, Fiori S, Guzzetta A, Perazza S, Sicola E, Cioni G. Spastic diplegia in preterm-born children: Executive function impairment and neuroanatomical correlates. Res Dev Disabil. 2017 Feb;61:116-126. doi: 10.1016/j.ridd.2016.12.006. Epub 2017 Jan 7. PMID 28073076
- [Background] Pirila S, van der Meere J, Korhonen P, Ruusu-Niemi P, Kyntaja M, Nieminen P, Korpela R. A retrospective neurocognitive study in children with spastic diplegia. Dev Neuropsychol. 2004;26(3):679-90. doi: 10.1207/s15326942dn2603_2. PMID 15525564
- [Background] Schatz J, Craft S, White D, Park TS, Figiel GS. Inhibition of return in children with perinatal brain injury. J Int Neuropsychol Soc. 2001 Mar;7(3):275-84. doi: 10.1017/s1355617701733012. PMID 11311028
- [Background] Bodimeade HL, Whittingham K, Lloyd O, Boyd RN. Executive function in children and adolescents with unilateral cerebral palsy. Dev Med Child Neurol. 2013 Oct;55(10):926-33. doi: 10.1111/dmcn.12195. Epub 2013 Jun 28. PMID 23809003
- [Background] Pirila S, van der Meere JJ, Rantanen K, Jokiluoma M, Eriksson K. Executive functions in youth with spastic cerebral palsy. J Child Neurol. 2011 Jul;26(7):817-21. doi: 10.1177/0883073810392584. Epub 2011 Mar 11. PMID 21398561
- [Background] Critten V, Messer D, Sheehy K. Delays in the reading and spelling of children with cerebral palsy: Associations with phonological and visual processes. Res Dev Disabil. 2019 Feb;85:131-142. doi: 10.1016/j.ridd.2018.12.001. Epub 2018 Dec 13. PMID 30553174
- [Background] Cantin RH, Gnaedinger EK, Gallaway KC, Hesson-McInnis MS, Hund AM. Executive functioning predicts reading, mathematics, and theory of mind during the elementary years. J Exp Child Psychol. 2016 Jun;146:66-78. doi: 10.1016/j.jecp.2016.01.014. Epub 2016 Feb 23. PMID 26914106
- [Background] Cartwright KB, Marshall TR, Huemer CM, Payne JB. Executive function in the classroom: Cognitive flexibility supports reading fluency for typical readers and teacher-identified low-achieving readers. Res Dev Disabil. 2019 May;88:42-52. doi: 10.1016/j.ridd.2019.01.011. Epub 2019 Mar 6. PMID 30851482
- [Background] Garcia-Galant M, Blasco M, Reid L, Pannek K, Leiva D, Laporta-Hoyos O, Ballester-Plane J, Miralbell J, Caldu X, Alonso X, Toro-Tamargo E, Melendez-Plumed M, Gimeno F, Coronas M, Soro-Camats E, Boyd R, Pueyo R. Study protocol of a randomized controlled trial of home-based computerized executive function training for children with cerebral palsy. BMC Pediatr. 2020 Jan 7;20(1):9. doi: 10.1186/s12887-019-1904-x. PMID 31910803
- [Background] Miyake A, Friedman NP, Emerson MJ, Witzki AH, Howerter A, Wager TD. The unity and diversity of executive functions and their contributions to complex "Frontal Lobe" tasks: a latent variable analysis. Cogn Psychol. 2000 Aug;41(1):49-100. doi: 10.1006/cogp.1999.0734. PMID 10945922
- [Background] Bombonato C, Del Lucchese B, Ruffini C, Di Lieto MC, Brovedani P, Sgandurra G, Cioni G, Pecini C. Far Transfer Effects of Trainings on Executive Functions in Neurodevelopmental Disorders: A Systematic Review and Metanalysis. Neuropsychol Rev. 2024 Mar;34(1):98-133. doi: 10.1007/s11065-022-09574-z. Epub 2023 Jan 12. PMID 36633797
- [Background] Ballester-Plane J, Laporta-Hoyos O, Macaya A, Poo P, Melendez-Plumed M, Toro-Tamargo E, Gimeno F, Narberhaus A, Segarra D, Pueyo R. Cognitive functioning in dyskinetic cerebral palsy: Its relation to motor function, communication and epilepsy. Eur J Paediatr Neurol. 2018 Jan;22(1):102-112. doi: 10.1016/j.ejpn.2017.10.006. Epub 2017 Oct 24. PMID 29108712
- [Background] Capodieci A, Romano M, Castro E, Di Lieto MC, Bonetti S, Spoglianti S, Pecini C. Executive Functions and Rapid Automatized Naming: A New Tele-Rehabilitation Approach in Children with Language and Learning Disorders. Children (Basel). 2022 Jun 2;9(6):822. doi: 10.3390/children9060822. PMID 35740759